CLINICAL TRIAL: NCT00374478
Title: Effects of Transdermal Scopolamine on Occupational Performance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CDC R49/CCR115279-5
Record Dates: First submitted 2006-02-02; First posted 2006-09-11 (Estimated); Last update posted 2007-04-09 (Estimated); Status verified 2007-04

CONDITIONS: Motion Sickness
Keywords: Scopolamine; Antiemetic; Task performance and analysis; Psychomotor vigilance test
MeSH Terms: conditions — Motion Sickness | interventions — Scopolamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Scopolamine

SUMMARY:
The purpose of this study is to determine the effects of Transdermal scopolamine vs. placebo on ship navigation performance under simulated heavy sea conditions.

DETAILED DESCRIPTION:
Our study proposes to use a randomized crossover placebo controlled design to test the effects of transdermal scopolamine vs. placebo on simulated ship navigation performance under conditions of heavy seas. We hypothesize that mariners will experience a greater decrement in navigational performance in the placebo condition vs. transdermal scopolamine, when faced with simulated heavy seas. Study staff will apply the transdermal scopolamine patch or placebo patch, 8 hours prior to performance assessment. Participants will surrender car keys and will agree stay on the Kalmar Maritime Campus until they are dismissed from the study. A study nurse and/or study physician will be on call from the time of patch application until study participants are dismissed from the study. Eight hours following patch application participants will perform navigation tasks, under stormy weather conditions, in the bridge simulation lab at Kalmar Maritime Academy. Participants will repeat the protocol one week later under the opposite dosing condition. This study will be conducted at the Kalmar Maritime Academy, Kalmar, Sweden.

ELIGIBILITY:
Inclusion Criteria:

* 20-60 years of age;
* English speaking;
* Marine cadets and officers with ship handling experience who volunteer for the study and agree to participate in ship simulation familiarization training prior to study commencement;
* Agree to refrain from alcohol use for 24 hours prior to dosing;
* Agree to stay on Kalmar Maritime Campus after scopolamine or placebo drug patch is applied and until study staff approves dismissal;
* Agree to remain at study site until passing sobriety test and dry mouth assessment;
* Agree to refrain from driving and operating heavy machinery after patch is applied and for 24 hours following patch removal;
* Agree to refrain from alcohol use 24 hours following patch removal at Sessions Two and Three;
* Agree to surrender car keys upon arrival at study site;
* Agree to receive a cab ride home from study;
* Females who are not pregnant as measured by a home pregnancy test prior to application of Transdermal scopolamine;
* Females who are using reliable birth control, per self report, not taking prescription or non prescription drugs contraindicated for Transdermal scopolamine use;
* Must weigh between 130 ( 58.9 7kgs)-260( 117.93 kgs) pounds;
* Must score less than a 5 on the Short Version- Michigan Alcohol Screening Test;
* No history of medical conditions contraindicated for Transdermal scopolamine use.

Exclusion Criteria:

* Individuals who are under 20 years of age or older than 60;
* Non-English speaking;
* Females who are pregnant (as measured by EPT pregnancy test prior to application of Transdermal scopolamine);
* Females who are not using reliable birth control, per to self report;
* A score of 5 or more on the SMAST (Short Version- Michigan Alcohol Screening Test);
* Reported use of recreational drugs;
* Reported history of treatment for alcohol or substance abuse;
* Currently taking prescription or non-prescription medications contraindicated for use with Transdermal scopolamine as per Physician's Desk Reference (including sedatives, tranquilizers, belladonna alkaloids, antihistamines, tricyclic antidepressants, and muscle relaxants);
* Reported history of medical conditions contraindicated for Transdermal scopolamine use (including pyloric obstruction, urinary bladder neck obstruction, impaired liver or kidney function, glaucoma, heart condition, obstructions to the stomach or intestines, prostrate enlargement, seizure history or psychosis);
* Participants weighing less than 130 lbs ( 58.9 7kg) and greater than 260( 117.93 kg);
* Allergic to adhesive materials; alcohol consumption 24 hours prior to dosing.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33
Dates: Start 2005-04; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
simulated ship navigation performance eight hours following Transdermal scopolamine application

SECONDARY OUTCOMES:
effectiveness of psychomotor vigilance testing as a fitness-for-duty test

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Howland, Ph.D., MPH, Principal Investigator — Boston University
Locations (1):
- Kalmar Maritime Academy, Kalmar, Sweden